# Evaluation of the New Veress Needle + Mechanism: A Pre-Clinical Study on Thiel Embalmed Bodies

## Principal Investigators:

- Roelf R Postema MD, consultant Surgeon, Amsterdam University Medical Centers, The Netherlands
- Tim Horeman MSc PhD, assistant Professor, University of Technology Delft, The Netherlands
- David Cefai MSc, Provinci Medtech, Nootdorp, The Netherlands
- Jean Calleja-Agius MD PhD, Professor of Gynecology, University of Malta, Malta

#### **Study Location:**

Laboratory for Anatomy, Biomedical Building, University of Malta, Msida, MSD2080 Malta

### Study dates:

20-24 September 2021

# Evaluation of the New Veress Needle + Mechanism: A Pre-Clinical Study on Thiel Embalmed Bodies

| | • |
|---|---|
| Nr: Participant's Consent Form | |
| | ndersigned, give my consent to take part in the study conducted by Provinci medtech, TU Delft and versity of Malta. This consent form specifies the terms of my participation in this research study. |
| 1. | I have been given written and/or verbal information about the purpose of the study; I have had the opportunity to ask questions and any questions that I had were answered fully and to my satisfaction. |
| 2. | I also understand that I am free to accept to participate, or to refuse or stop participation at any time without giving any reason and without any penalty. Should I choose to participate, I may choose to decline to answer any questions asked. In the event that I choose to withdraw from the study, any data collected from me will be erased as long as this is technically possible (for example, before it is anonymised or published), unless erasure of data would render impossible or seriously impair achievement of the research objectives, in which case it shall be retained in an anonymised form. |
| 3. | I understand that I have been invited to participate in one clinical study. |
| 4. | I understand that, under the General Data Protection Regulation (GDPR) and national legislation, I have the right to access, rectify, and where applicable, ask for the data concerning me to be erased. |
| 5. | I understand that all data collected will be stored in an anonymised form |
| 6. | I am aware that I am giving my consent to be video recorded where said video material can only be used when anonymised. |
| | I have read and understood the above statements and agree to participate in this study. |
| | Name of participant: |
| | Signature: |